CLINICAL TRIAL: NCT07404748
Title: The Effect of Stress Management Training on Perceived Stress and Life Satisfaction: An Experimental Mediation Analysis
Brief Title: Stress Management and Life Satisfaction in University Students
Acronym: USSMLS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Erzincan Binali Yildirim Universitesi (Other)
Responsible Party: Principal Investigator, Feyza KARSLI, Assistant Professor, Erzincan Binali Yildirim Universitesi
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: Protocol No: 11/03
Record Dates: First submitted 2025-12-19; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Stress Management; Coping Skills; Youth Mental Health
Keywords: Psychoeducation; Stress management; Coping skills; Young adults; Youth mental health

STUDY DESIGN:
Intervention Model Description: This study employs a 2×2 factorial randomized design. Participants are randomly assigned to four groups based on the presence or absence of the intervention component and the presence or absence of the stress task. This design allows for the examination of the main and interaction effects of the intervention components.
Masking Description: Not applicable. This is an open-label study with no masking.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control Group (No Stress Education, No Stress Task) (No Intervention): Participants in this group receive neither stress training nor stress tasks.
- Stress Task Only (No Stress Education) (Experimental): Participants in this group receive stress-related tasks that do not involve stress training.
  Interventions: Behavioral: Stress Task
- Stress Education Only (No Stress Task) (Experimental): Participants in this group receive stress training without any stressful tasks.
  Interventions: Behavioral: Stress Education
- Stress Education + Stress Task (Experimental): Participants in this group receive both stress training and the task.
  Interventions: Behavioral: Stress Education; Behavioral: Stress Task

INTERVENTIONS:
Behavioral: Stress Education — A structured stress training program designed to increase participants' awareness of stress and teach them basic stress management and coping strategies.
  Arms: Stress Education + Stress Task; Stress Education Only (No Stress Task)
Behavioral: Stress Task — A stress task-based intervention that includes structured activities designed to engage participants and encourage active participation.
  Arms: Stress Education + Stress Task; Stress Task Only (No Stress Education)

SUMMARY:
This study aims to examine the effects of a structured psychoeducational program on the psychological well-being of university students. Participants will be randomly assigned to either a psychoeducational group or a control group. The psychoeducational program includes sessions designed to improve stress coping skills. Data will be collected using self-report questionnaires administered after the intervention. The study does not involve any drugs or medical devices and is considered to be of minimal risk. The findings are expected to contribute to the development of effective psychosocial interventions for young adults.

DETAILED DESCRIPTION:
This study is designed to evaluate the relationship between coping with stress, perceived stress, and life satisfaction within a causal framework using an experimental mediating model. The study examines the effect of structured stress coping training on participants' perceived stress and life satisfaction. Psychoeducation is widely used in mental health settings to improve individuals' understanding of emotions, stress, and coping strategies. However, evidence regarding its effectiveness in specific populations is limited. Participants will be randomly assigned to either an intervention group receiving a psychoeducation program and performing a stress task, or a control group receiving no intervention and performing a stress task, for the duration of the study. The psychoeducation program will be delivered in a group format and will focus on topics such as emotional awareness, stress management, adaptive coping skills, and problem-solving. Data will be collected using self-report measures following completion of the intervention. The study does not involve any pharmacological treatment or medical devices and is considered to be of minimal risk. The results of this study are expected to shed light on future psychosocial intervention programs.

ELIGIBILITY:
Inclusion Criteria:

* Being a university student
* Willingness to participate voluntarily in the study
* Attendance at all sessions throughout the education program
* No prior participation in a similar stress management or stress coping education program

Exclusion Criteria:

* Not being a university student
* Not providing voluntary consent to participate in the study
* Irregular attendance or non-completion of the education sessions
* Previous participation in a similar stress management or stress coping education program

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-02-16 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Life Satisfaction Score (Satisfaction With Life Scale) | Baseline and 4 weeks
  Life satisfaction was assessed using the Satisfaction With Life Scale (SWLS) developed by Diener et al. (1985), a validated self-report measure. The scale consists of 5 items rated on a 7-point Likert scale, yielding total scores ranging from 5 to 35. Higher scores indicate greater life satisfaction.

SECONDARY OUTCOMES:
Perceived Stress Score (Perceived Stress Scale-14) | Baseline and 4 weeks
  Perceived stress was assessed using the Perceived Stress Scale-14 (PSS-14) developed by Cohen, Kamarck, and Mermelstein (1983), a validated self-report questionnaire designed to measure the degree to which situations in one's life are appraised as stressful. The scale consists of 14 items rated on a 5-point Likert scale ranging from 0 (never) to 4 (very often). Total scores range from 0 to 56, with higher scores indicating greater perceived stress. Seven positively stated items are reverse scored.

CONTACTS AND LOCATIONS:
Overall Officials: FEYZA KARSLI, Principal Investigator — Erzincan Binali Yıldırım University, Department of Psychology

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared due to ethical and confidentiality considerations, as the study involves sensitive psychological information and participants did not provide consent for data sharing.